CLINICAL TRIAL: NCT06174675
Title: Combined Bilateral Infraorbital and Infratrochlear Nerve Block Versus Conventional Systemic Analgesia for Patients Undergoing Nasal Surgeries
Brief Title: The Effect of Combined Bilateral Infraorbital and Infratrochlear Nerve Block in Nasal Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ayat Mohamed Elshaer, assistant lecturer of anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FMASU MD136/2023
Record Dates: First submitted 2023-12-08; First posted 2023-12-18 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Active Comparator): patients will receive combined bilateral infraorbital and infratrochlear nerve block.
  20 patients
  Interventions: Procedure: combined bilateral infraorbital and infratrochlear nerve blocks
- control group (No Intervention): patients will not receive the block and will receive intravenous analgesia according to standard protocol.
  20 patients.

INTERVENTIONS:
Procedure: combined bilateral infraorbital and infratrochlear nerve blocks — Filling the block labelled syringe with 8 mL of bupivacaine 0.25%. Starting with Infraorbital nerve block using an extraoral approach.Inserting a 25-gauge needle laterally to the ipsilateral nostril after palpating the infraorbital ridge to locate the infraorbital foramen. Positioning of the index finger of the non-dominant hand above the infraorbital foramen and advancing the needle feeling it beneath the finger to avoid globe penetration injury. Injecting 3 mL of the study solution slowly after confirming negative aspiration of blood and taking care not to inject into the foramen itself.
  Shifting to infratrochlear nerve block by inserting the needle 1 cm above the inner canthus targeting the junction of the orbit and the nasal bone. Injecting 1mL of the study solution after confirming negative aspiration of blood.
  Performing contralateral nerve block in the same manner. Applying pressure to four injection points for one minute to prevent hematoma.
  Arms: Study group

SUMMARY:
The aim of the study is to assess the efficacy of adding a pre-emptive combined bilateral infraorbital and infratrochlear nerve blocks with bupivacaine 0.25% in decreasing intraoperative and postoperative analgesics consumption and maintaining intraoperative hemodynamic stability during nasal surgeries.

DETAILED DESCRIPTION:
Perioperative pain management is one of the most important issues of most surgical procedures. The goal of every pain management technique is to reduce or eliminate pain and discomfort with minimum side effects (Garmella and Cellini, 2012).

Nasal surgical procedures are associated with a high incidence of emergence agitation leading to severe complications such as bleeding and delayed recovery which increase the hospital stay (Kim et al., 2015).

Although the cause of emergence agitation is not well established, Pain in the immediate post-operative period is one of the significant risk factors for emergence agitation. Multiple analgesic interventions are applied to the patient before, during and after surgery prevent these complications (Gray et al., 2018).

The most utilized analgesic interventions are combinations of narcotic and non-steroidal anti-inflammatory drugs. However, they are associated with gastrointestinal and neurological side effects which cause discomfort to the patient and affect surgical recovery profile (Çelik et al., 2018). Therefore, the utility of combining regional nerve block with general anesthesia has been popularized in clinical practice to provide improved perioperative analgesia, decreased narcotic consumption and enhanced emergence and recovery characteristics (Mariano et al., 2009; Ibrahim et al., 2018).

The infraorbital nerve (ION) is a branch of the maxillary part of the trigeminal nerve. This nerve innervates the skin of the nose and septum mobile nasi. The infratrochlear nerve (ITN) innervates the root of the nose and is an extraconal branch of the nasociliary nerve, which is a branch of the ophthalmic portion of the trigeminal nerve (Choi et al., 2019).

Although these nerve blocks are simple and easy to use with few complications, there are limited reports that suggest combined bilateral infraorbital and infratrochlear nerve blocks to be effective to facilitate pain management and reduce anesthetic agent consumption and perioperative dose of narcotics in nasal procedures (Cekic et al., 2013; Boselli et al., 2016).

ELIGIBILITY:
Inclusion Criteria:

1. Age group: 18 - 55 years old.
2. American Society of Anesthesiologists (ASA) Physical Status Class I or II
3. Scheduled for elective nasal surgery under general anesthesia.

Exclusion Criteria:

1. Refusing to participate in the study or inability to provide informed consent.
2. History of allergy to the medications used in the study.
3. Contraindications to regional anesthesia (including coagulopathy, INR ≥ 1.4 and local infection).
4. Compromised renal or liver functions.
5. History of substance or alcohol abuse.
6. Pre-existing chronic pain of different etiology.
7. Psychiatric disorders.
8. Pregnancy.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
Total amount of intraoperative fentanyl | throughout the surgery

SECONDARY OUTCOMES:
1. Hemodynamic changes | every 15 minutes during the surgery, upon arrival to the PACU and after 30 min.
  mean arterial blood pressure (MAP), heart rate (HR) will be recorded before anesthesia,
The time from induction of anesthesia to the first additional dose of fentanyl intraoperative. | throughout the surgery
Total amount of postoperative pethidine given | 24 hours postoperatively
Number of patients needed rescue analgesia intraoperative or postoperative. | throughout the surgery and 24 hours postoperatively
Any complications related to the nerve block such as injection site pain, edema, hematoma or neurological deficits in the blocked area such as paresthesia or prolonged paralysis of the upper lip. | 24 hours postoperatively
Postoperative side effects such as nausea, vomiting and headache. | 24 hours postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Ayat Elshaer, ass.lecturer, Principal Investigator — faculty of medicine, Ain Shams University
Locations (1):
- Ain shams university hospitals, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No